CLINICAL TRIAL: NCT06141057
Title: Phase I Clinical Trial to Assess the Safety and Immunogenicity of the Malaria Vaccine Candidate RH5.1 Soluble Protein in Matrix-MTM Using Two Dosing Regimens
Brief Title: A Study to Compare Two Dosing Regimens for a New Malaria Vaccine
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-002
Record Dates: First submitted 2023-07-14; First posted 2023-11-21 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Malaria; Malaria,Falciparum; Protozoan Infections; Parasitic Disease; Infections; Vector Borne Diseases
Keywords: RH5.1; Matrix-M
MeSH Terms: conditions — Malaria; Malaria, Falciparum; Protozoan Infections; Parasitic Diseases; Infections; Vector Borne Diseases | interventions — Matrix-M

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Delayed regimen (Experimental): 12 volunteers receiving three doses of 10 µg RH5.1 with 50 µg of Matrix-M on days 0, 28 and 182 via intramuscular (IM) injection in the deltoid region of the non-dominant arm
  Interventions: Biological: Matrix M with RH5.1
- Group 2: Delayed Fractional Regimen (Experimental): 12 volunteers receiving two doses of 50 µg RH5.1 with 50 µg of Matrix-M on days 0, 28 and one dose of 10 µg RH5.1 with 50 µg of Matrix-M on day 182 via intramuscular (IM) injection in the deltoid region of the non-dominant arm
  Interventions: Biological: Matrix M with RH5.1

INTERVENTIONS:
Biological: Matrix M with RH5.1 — 50 µg of Matrix-M adjuvant with RH5.1 at different doses on days 0 and 28.

SUMMARY:
Malaria is a major public health problem. There were around 240 million cases of malaria and 627,000 deaths worldwide in 2020. Most of the deaths are in children under five living in Africa. It is a major problem for those who live in affected areas and for travellers. There is a great need for a safe, effective malaria vaccine.

This study is being done to evaluate an experimental malaria vaccine for its safety and also look at the body's immune response to the vaccine.

The vaccine tested in this study is called and "RH5.1". This is given with an adjuvant called "Matrix-M". This is a substance to improve the body's response to a vaccination.

The aim is to use the vaccines and adjuvant to help the body make an immune response against parts of the malaria parasite. This study will assess:

1. The safety of the vaccines in healthy participants.
2. The response of the human immune system to the vaccines.

This will be achieved by giving participants three doses of the RH5.1 vaccines at two different dose levels (10 micrograms and 50 micrograms). One group will have 3 doses of 10 micrograms given at 0, 1 and 6 months whilst the other will receive 2 doses of 50 micrograms (at 1 and 2 months) followed by a 10 microgram dose at 6 months- known as a 'delayed fractional dose'. Blood tests and information about any symptoms will be performed/collected that occur after vaccination.

Information from previous studies suggests that a delayed fractional dose improves the immune response to the vaccine, particularly in terms of the antibody response. Current prediction is that this improvement is due to the delay in dosing, rather than the reduction in dose, and this study will help to answer that. Having a vaccine at a single dose is important for efficient production and dosing for vaccines rolled out in national programs so being able to move away from 'delayed fractional dose' regimens to 'delayed final dose' regimens will be important for vaccine development.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the Investigators to discuss the volunteer's medical history with their GP
* Participants of childbearing potential only: must practice continuous effective contraception for the duration of the study (see section 9.9)
* Agreement to refrain from blood donation for the duration of the study
* Able and willing to provide written informed consent to participate in the trial

Exclusion Criteria:

* History of clinical malaria (any species) or previous participation in any malaria (vaccine) trial or controlled human malaria infection (CHMI) study
* Travel to a clearly malaria endemic locality during the study period or within the preceding six months
* Use of immunoglobulins or blood products (e.g. blood transfusion) in the last three months
* Receipt of any vaccine in the 30 days preceding enrolment, or planned receipt of any other vaccine within 30 days following each study vaccination, with the exception of COVID-19 vaccines, which should not be received between 14 days before to 7 days after any study vaccination
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period
* Concurrent involvement in another clinical trial involving an investigational product or planned involvement during the study period
* Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data, as assessed by the Investigator
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
* Any history of anaphylaxis
* Pregnancy, lactation or intention to become pregnant during the study
* Body mass index of <18.5 or >35
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition that may affect participation in the study
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol misuse as defined by an alcohol intake of greater than 25 standard UK units every week
* Suspected or known injecting drug use in the 5 years preceding enrolment
* Hepatitis B surface antigen (HBsAg) detected in serum
* Seropositive for hepatitis C virus (antibodies to HCV) at screening (unless volunteer has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV ribonucleic acid (RNA) PCR at screening for this study)
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination. Blood test abnormalities will be assessed as per the laboratory adverse event table in Appendix A (table 8). In the event of abnormal test results deemed to be clinically significant, confirmatory repeat tests may be requested. Procedures for identifying laboratory values meeting exclusion criteria are described in Appendix A.
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of RH5.1 soluble protein in Matrix-M in healthy adult volunteers by assessing the occurrence of solicited reactogenicity following each vaccinations | 7 days following each vaccination
  Occurrence of solicited local/systemic reactogenicity signs and symptoms for 7 days. following each vaccination. These will be tabulated, detailing frequency, duration and severity of signs and symptoms.
To assess the safety of RH5.1 soluble protein in Matrix-M in healthy adult volunteers by assessing the occurrence of unsolicited adverse events following each vaccinations | 28 days following each vaccination
  Occurrence of unsolicited adverse events for 28 days following the vaccination. These will be tabulated, detailing frequency, duration and severity of AEs.
To assess the safety of RH5.1 soluble protein in Matrix-M in healthy adult volunteers by comparing safety laboratory measures following each vaccinations | 28 days following each vaccination
  Change from baseline for safety laboratory measures for 28 days following vaccination. Haematological and biochemical laboratory values will be presented according to local grading scales.
To assess the safety of RH5.1 soluble protein in Matrix-M in healthy adult volunteers by assessing the occurrence of serious adverse events | During Whole study duration (547 days)
  Occurrence of serious adverse events during the whole study duration. These will be tabulated, detailing frequency, duration and severity of SAEs.

SECONDARY OUTCOMES:
To assess the humoral immunogenicity of RH5.1 soluble protein with Matrix-M when administered to healthy volunteers at different doses. | From a number of key timepoints (Baseline up to day 547)
  Serum ELISA response, quantitative antigen-specific IgG antibody levels (µg/mL readout) over time - analysis of peak responses and longevity, with comparison before and after vaccination
To compare the anti-RH5 serum IgG functional immunogenicity between the two groups receiving soluble RH5.1 at different doses by assessing purified IgG versus GIA titration (quality analysis) | After each vaccinations (D0, D28 and D182)
  Immunogenicity will be assessed to characterise quantity, quality and longevity of serum anti-RH5 IgG responses as measured by standardised ELISA. The growth inhibition activity will be used to determine functionality of these responses and allow quality analysis. Comparisons between two groups receiving soluble RH5.1 protein at different doses will be made post vaccination to determine how differing doses affect these responses.
To compare differences in the innate immune responses following the first and third vaccinations and correlated these with adverse event data and adaptive immune responses | 7, 28 days following first and third vaccinations
  Innate immune cell analyses will include flow cytometry analyses and quantitative measurements of pro-inflammatory cytokines to phenotype innate immune cell populations primarily in the first 7 days following vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals, Royal Hallamshire Hospital, Sheffield, United Kingdom